CLINICAL TRIAL: NCT04378296
Title: Economic Evaluation in Dermatology: Teledermatology Versus Conventional Monitoring of Patients in the Hospital
Brief Title: Economic Evaluation in Teledermatology
Acronym: TELEDERMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antonio Lopez Villegas (Other)
Collaborators: Universidad de Almeria (Other)
Responsible Party: Sponsor-Investigator, Antonio Lopez Villegas, Principal Investigator, Universidad de Almeria
Organization: Universidad de Almeria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 27/2020; PI_20_12CS Telederma (Registry Identifier: Hospital de Poniente)
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Skin Diseases
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teledermatology (Experimental): The 221 patients who are included in this group will be monitored from the Primary Care centers.
  Interventions: Other: Teledermatology
- Conventional monitoring (No Intervention): The 221 patients included in this group will have to visit the dermatologist at the hospital.

INTERVENTIONS:
Other: Teledermatology — The experimental group will be made up of dermatological patients monitored asynchronously.
  Arms: Teledermatology

SUMMARY:
Introduction: Previous studies confirm that teledermatology allows the generation of a quick response from the specialist's consultation, reduction of unnecessary travels, early diagnosis and priority in the attention to the most urgent cases. Despite these advantages and that teledermatology has experienced exponential growth since its introduction approximately 16 years ago in Spain, in Andalusia, its use is still very limited. The objective of this project will be to carry out an analysis of the quality of life related to health, costs, cost-utility and informal care of teledermatology services in Primary Care compared to conventional monitoring carried out at the Hospital de Poniente.

Methodology: A randomized, controlled, unmasked, inter-level clinical trial (Primary Care-Hospital de Poniente) and multicentre (all health centers attached to the Poniente Health District of Almería) will be carried out with a 6-month follow-up. Patients will be assigned to the teledermatology group (experimental) or the conventional monitoring group in the hospital (control). The patients included in the experimental group will be monitored asynchronously. Baseline characteristics, number of visits to the hospital, health-related quality of life, costs, informal care and satisfaction from the perspective of the Andalusian Public Health System and patients and their caregivers will be analyzed. The generic EuroQol-5D questionnaire (EQ-5D) will be administered to assess health-related quality of life and the SKINDEX-29 quality of life dermatological questionnaire. A cost-utility analysis will be performed to assess whether tele-dermatology is cost-effective in terms of additional cost for additional quality-adjusted life years (QALYs).

ELIGIBILITY:
Inclusion Criteria:

* 1. Be over 18 years old.
* 2. Having any skin disease.
* 3. Accept to participate in the study.

Exclusion Criteria:

* 1. Non-dermatological disease.
* 2. Be participating in another study.
* 3. Refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
EuroQol-5Dimensions questionnaire | 6 months
  From -1 [the poorest imaginable health state] to 1 [perfect health]

SECONDARY OUTCOMES:
Clinical features | 6 months
  Patient's age; sex; diagnosis; origin; indication (type of dermatological problem); number of visits
Dermatological Quality of Life Questionnaire | 6 months
  0 (no effect on quality of life) up to 100 (maximum effect on quality of life)
Healthcare costs | 6 months
  Costs paid by the Public Health System
Informal cost | 6 months
  Costs paid by the patients
In-depth interviews on the healthcare received in Primary Care centers | 6 months
  1) healthcare center, 2) procedure to make an appointment, 3) medical consultation, 4) nursing consultation
Health Care Communication Questionnaire | 6 months
  The 5-point Likert scale, ranging from 1 (not at all) to 5 (very much).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lopez-Villegas, PhD, Principal Investigator — Hospital de Poniente
Locations (2):
- Spain (2):
  - Hospital de Poniente, El Ejido, Almeria
  - Antonio López-Villegas, El Ejido, Almería